CLINICAL TRIAL: NCT00976365
Title: Phase IIa Study of Metastatic Breast Cancer
Brief Title: Evaluation of the Safety and Efficacy of THL-P in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan THL Co.LTd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: King-Jen Chang, / Surgy, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THL-P; NTUH-REC No.2008100025M
Record Dates: First submitted 2009-07-06; First posted 2009-09-14 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THL-P (Experimental): Solution for study only.
  Interventions: Dietary Supplement: THL-P
- Sugar pill (Placebo Comparator): THL-p
  Interventions: Dietary Supplement: THL-P

INTERVENTIONS:
Dietary Supplement: THL-P — 20ml/bottle, TID, 24weeks
  Other Names: THL-P solution

SUMMARY:
The purpose of this study is to obtain evidence from test article with efficacy in Metastatic Breast Cancer patients. The average of all changes from baseline to post-treatment evaluations in global health/quality of life (QoL) subscale assessed by self-administered European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC-QLQ-C30).

DETAILED DESCRIPTION:
The test article is extracted from many natural herbals, in which most or their components have been shown to have anti-tumor activity. A study in 2004 showed the test article could have strong immunomodulatory effect on the antigen-stimulated proliferation response (PR) of peripheral blood mononuclear cells (PBMC) and T-cells from recurrent aphthous ulcerations (RAU) patients and suggested that it might be a potential immunoceutical agent for treatment of RAU. Subsequent study in 2005 also suggested the test article as a potential immunoceutical agent for treatment of RAU because the result showed it could modulate the antigen-stimulated cytokine production by T-cells isolated from RAU patients. Another study in 2005 showed the test article also had a broad-range tumor killing function and provided a molecular basis underlying therapeutic activity. It was also suggested in this study will could be a potential and promising cancer therapeutic or preventive agent.

The aim of this current study is to explore the safety and efficacy of the investigational product with 20 ml, 3 times per day (daily dose: 60 ml) for a total of 24 weeks in the patients with metastatic breast cancer refractory to conventional treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed breast cancer with clinical evidence.
* Life expectancy of at least 4 weeks.

Exclusion Criteria:

* Any Uncontrolled infection.
* Lupus erythematosus.
* Malignant tumor.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
QOL | 6 months measure

SECONDARY OUTCOMES:
CBC with platelet and differential counts. AST, ALT, total bilirubin, BUN, uric acid and Creatinine | 6 months measure

CONTACTS AND LOCATIONS:
Overall Officials: King-Jen Chang, M.D.,Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan